CLINICAL TRIAL: NCT04846530
Title: A Prospective, Single Blind, Single-center Study Evaluating the Histology and Intradermal Implantation of the Teosyal RHA® Collection of Fillers
Brief Title: Teosyal RHA® Histology and Intradermal Implantation Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2030403
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Histology
Keywords: Histology

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Approved products will be placed in small boluses (0.2 mL) intradermally: Subjects will be assigned to receive two products each from the RHA® line of products (RHA® 1, RHA® 2, RHA® 3, and RHA® 4).
  Interventions: Device: RHA® 1, RHA® 2, RHA® 3, and RHA® 4

INTERVENTIONS:
Device: RHA® 1, RHA® 2, RHA® 3, and RHA® 4 — For each subject, two spaced boluses (0.2 mL each) of the product will be implanted on the same side (left or right side) in the post auricular area of the subject per treatment assignment. The assignment will specify one of the RHA® products to the left ear and another product to the right ear. Each subject will have a total of four boluses.

SUMMARY:
The Teosyal RHA® family of products (RHA® 1, RHA® 2, RHA® 3, and RHA® 4) is approved in Canada for the correction of facial wrinkles and folds. In this study, the approved products will be placed in small boluses (0.2 mL) intradermally to allow for punch biopsies of the post-auricular space to be taken. The biopsies will include the injected material and surrounding skin tissue. Biopsies will be taken immediately after implantation of the product and at Day 30 and assessed by an independent blinded pathologist.

ELIGIBILITY:
Inclusion Criteria:

* 1. Outpatient, male or non-pregnant, non-nursing females, at least 22 years of age, and in good general health.

  2. Subject willing to abstain from other aesthetic procedures on the head or face including receiving other dermal fillers, laser treatments, use of any product that affects skin remodeling, or a product that may cause an active dermal response in the treatment area from screening through the last study follow-up visit.

  3. Female subjects of childbearing potential must have a negative urine pregnancy test result at the Treatment Visit, prior to product administration.

  4. Able to understand the requirements of the trial and sign informed consent including authorization to release health information.

  5. Subject willing and able to comply with study follow-up procedures and schedule.

  6. Subject willing to provide written informed consent for their participation in the study including authorization to release health information.

Exclusion Criteria:

* 1. Subject is a female of childbearing potential (e.g., not postmenopausal for at least one year or has not had a hysterectomy or tubal ligation) not using medically effective birth control (e.g., hormonal methods such as birth control pills; implants; Intrauterine Device (IUDs), etc., in use at least 30 days prior to injection or barrier methods such as condom and spermicide in use at least 14 days prior to injection), or is pregnant, lactating, or plans to become pregnant during the study.

  2. Subject has participated in a clinical study in which an investigational device or drug was received in the 30 days prior to screening or plans to enroll in such a study during the course of the current study.

  3. Subject is an employee or direct relative of an employee of the investigational site or Sponsor.

  4. Subject has a serious or progressive disease, which, in the investigator's judgment, puts the subject at undue risk (e.g., uncontrolled diabetes, autoimmune pathology, cardiac pathologies).

  5. Subject has a local acute inflammatory process or infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events.

  6. Subject has a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.

  7. Subject has had an active skin disease in the treatment area within the past 6 months.

  8. Subject has scars, infection, rosacea, herpes, acne, blotches or other pathology behind the ears. Subject is predisposed to keloidosis or hypertrophic scarring.

  9. Subject has known allergy to hyaluronic acid, 1,4-butanediol diglycidyl ether (BDDE), gram-positive bacterial proteins or streptococcal proteins.

  10. Subject has history of hypersensitivity to local anesthetics of the amide type, such as lidocaine.

  11. Subject has severe allergies as manifested by a history of anaphylaxis, or a history or presence of multiple severe allergies.

  12. Subject has a known bleeding disorder. 13. Subject has received or plans to receive within 1 week prior to injection through 1 week following or in the one week prior to 30 day biopsy through 1 week after any treatment/procedure that may impact coagulation such as high-dose Vitamin E, aspirin, anti-inflammatories, antiplatelets, thrombolytics, or any other medication that could increase the risk of bleeding. Subject has received within the past 3 months or plans to receive during the study chemotherapy agents, immunosuppressive medications, or systemic corticosteroids (inhaled steroids are acceptable).

  14. Subject has received within the past 12 months or plans to receive during the study any treatment or procedure involving the post-auricular area.

  15. Any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the trial results, or may interfere significantly with the subject's participation in the trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All healthy subjects who fulfill the entry criteria (inclusion and exclusion) will be considered for study recruitment.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
Biopsy specimens | Day 1
  The biopsy specimens will be submitted to an independent laboratory for histological examination.

SECONDARY OUTCOMES:
Biopsy specimens | Day 30
  The biopsy specimens will be submitted to an independent laboratory for histological examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Woodbridge, Ontario Site, Woodbridge, Ontario, Canada